CLINICAL TRIAL: NCT00120744
Title: Randomized Trial of the Oral Disintegrating Ondansetron Tablet to Reduce Vomiting From Acute Gastroenteritis in a Pediatric Emergency Department
Brief Title: Oral Disintegrating Ondansetron Tablet to Reduce Vomiting From Gastroenteritis in a Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); GlaxoSmithKline (Industry); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Stephen Freedman, Adjunct Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2003-12038
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Gastroenteritis; Vomiting; Diarrhea; Dehydration
MeSH Terms: conditions — Gastroenteritis; Vomiting; Diarrhea; Dehydration

INTERVENTIONS:
Drug: Ondansetron Oral Disintegrating Tablet

SUMMARY:
The objectives of the study were to determine whether ondansetron treatment would reduce:

* the amount of vomiting in the emergency department;
* the need for intravenous rehydration; and
* the need for hospitalization.

DETAILED DESCRIPTION:
Background:

Vomiting may limit the success of oral rehydration in children with gastroenteritis and dehydration. Limited data suggest that while oral ondansetron may reduce vomiting from gastroenteritis, emergency department revisits may increase.

Methods:

The investigators conducted a prospective, double-blind randomized trial at a pediatric emergency department in 214 dehydrated children, aged 6 months to 10 years with gastroenteritis and mild to moderate dehydration as assessed by a dehydration score. They were randomly assigned to receive treatment with an ondansetron oral disintegrating tablet or placebo. Oral rehydration was administered according to a standard protocol. The primary outcome was the proportion of children who vomited during oral rehydration therapy. The secondary outcomes were the mean number of episodes of vomiting, and the proportion of children treated with intravenous rehydration or hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Acute gastroenteritis
* Non-bilious and non-bloody vomiting within 4 hours of triage
* Diarrhea
* Mild to moderate dehydration

Exclusion Criteria:

* Weight less than 8 kilograms
* Severe dehydration
* Underlying disease which might affect the assessment of hydration status (e.g., chronic renal failure, hypoalbuminemia, congestive heart failure, on diuretics)
* History of abdominal surgery
* Hypersensitivity to the drug or any components in its formulation

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The proportion of children who vomit during oral rehydration therapy after receiving either 0.13-0.27 mg per kilogram of an oral disintegrating ondansetron tablet or placebo.

SECONDARY OUTCOMES:
To compare in each treatment arm: mean number of episodes of vomiting, the proportion of children administered supplemental intravenous rehydration or requiring hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Freedman, MDCM, MSCI, Principal Investigator — The Hospital for Sick Children